CLINICAL TRIAL: NCT02157025
Title: A More Engaging Visual Field Test to Increase Use and Reliability in Pediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KID_VF
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Suspect; Optic Nerve Hypoplasia and Abnormalities of the Central Nervous System; Congenital Coloboma of the Optic Nerve; Optic Nerve Head Pits, Bilateral Congenital
Keywords: Humphrey visual fields; perimetry; pediatrics
MeSH Terms: conditions — Ocular Hypertension; Optic Nerve Hypoplasia and Abnormalities of the Central Nervous System; Coloboma of optic nerve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cartoon Intervention (Experimental): Cartoon video fixation target and cartoon character voice audio instructions during Humphrey perimetry
  Interventions: Device: Cartoon video fixation target and cartoon character voice audio instructions during Humphrey perimetry
- Usual Care (Active Comparator): Usual care procedures for Humphrey perimetry in young children
  Interventions: Other: Usual Care procedures during Humphrey perimetry for children

INTERVENTIONS:
Device: Cartoon video fixation target and cartoon character voice audio instructions during Humphrey perimetry
  Arms: Cartoon Intervention
Other: Usual Care procedures during Humphrey perimetry for children
  Arms: Usual Care

SUMMARY:
The majority of young children do not think that visual field (VF) testing of peripheral vision is similar to a game; therefore, it is not surprising that they have difficulty maintaining attention during VF testing and thus the test reliability suffers as a consequence. Poor VF reliability has been a longstanding, major issue since it leads to an increased number of tests and/or longer duration of time needed to determine when there are true vision losses. Providers are less likely to obtain VF tests in children since the results are of doubtful value and challenging to interpret when they are inconsistent. Effectively this means that children with untreated, slowly progressive eye diseases may go undiagnosed and incur greater visual losses. The investigators aim to create a prototype device that the investigators hypothesize will make VF testing more engaging for young children, thus increasing their attention and consistency of their responses to the test stimuli, which in turn should improve VF reliability. The components include a microdisplay video screen (1.5" diameter) as the fixation target (instead of the standard LED light) displaying video clips of popular cartoon characters, and audio clips of impersonated cartoon character voices presented by the test operator to provide instructional feedback based on the child's performance during testing. Improved VF reliability from the investigators intervention would translate to improved diagnosis and care for young childrens' peripheral vision loss through widespread implementation of the investigators innovative, affordable and readily adoptable system at eye care providers' offices.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-8
* Seen previously in the clinics at Nova Southeastern University's The Eye Care Institute with a diagnosis for glaucoma suspect or optic nerve abnormalities
* Able and willing to complete VF testing at 2 study visits about a week apart
* Provide informed consent

Exclusion Criteria:

* History of having previously completed a VF test using Humphrey static perimetry
* Inability to understand study or communicate responses (cognitive impairment)
* Unable to understand, read and speak English fluently

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Humphrey Visual Field Test-Retest Variability of Mean Deviation scores (dB) | 1 week
  Within subject, the investigators will determine the coefficient of variation in the mean deviation scores obtained at the two sessions a week apart (dB). The investigators will test for significant differences between subjects who receive the intervention versus the usual care control group for the test-retest variability.

SECONDARY OUTCOMES:
Humphrey Visual Field Reliability Indices and Ratings | 1 week
  The investigators will test for significant differences between subjects who receive the intervention versus the usual care control group for the visual field reliability criteria (false negatives, false positives and fixation losses; expressed as %), and operator ratings (subjects' fixation, cooperation and fatigue; scale 1 to 5).

CONTACTS AND LOCATIONS:
Overall Officials: Ava Bittner, Study Director — University of California, Los Angeles
Locations (1):
- The Eye Care Institute, Fort Lauderdale, Florida, United States